CLINICAL TRIAL: NCT04274348
Title: Role of Staphylococci on Cytokine and T Cell Profiles in the Pathogenesis of Atopic Dermatitis and Eczema Herpeticum
Brief Title: Staphylococcal Toxins in Atopic Dermatitis and Eczema Herpeticum
Acronym: STADEH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-A01904-53
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis; Staphylococcus Aureus; Bacterial Toxins; Immune Response; Cytokines; T Cells Subsets
MeSH Terms: conditions — Dermatitis, Atopic; Staphylococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin biopsies and blood samples (Other)
  Interventions: Other: Skin biopsies and blood samples

INTERVENTIONS:
Other: Skin biopsies and blood samples — Two skin biopsies and 30 ml of blood will be collected.

SUMMARY:
Atopic dermatitis (AD) is the most common chronic inflammatory skin disease. Clinical studies have demonstrated a link between staphylococcal skin colonization and the pathogenesis of AD, but the implication of bacterial virulence factors remains largely uncharacterized. Finally, AD is often associated with herpes simplex skin infections. The aim of this project is to investigate the role of staphylococcal toxins in the exacerbation and maintenance of atopic skin inflammation and in the occurrence of infectious complications such as eczema herpeticum.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate AD (SCORAD between 25 and 50) or severe AD (SCORAD> 50)
* Skin lesions in the forearms
* Free subject, without neither guardianship, wardship nor subordination
* Patient with Social Security
* Informed and signed consent by the patient after clear and loyal information on the study

Exclusion Criteria:

* Age < 18 year-old
* Patients with mild AD (SCORAD < 25)
* Patients without skin lesions in the forearms
* Patients treated with dermocorticoid or calcineurin inhibitor for less than two weeks
* Patients under systemic treatment : Methotrexate, Ciclosporin, Mycophenolate Mofetil, Azathioprine, general corticosteroids for less than 4 weeks
* Patients under biological treatment : Dupilumab for less than 5 half-lives
* Patient without Social Security
* Pregnant and nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Quantification of S. aureus colonization level and characterization of bacterial virulence profile in AD lesions. | 2 hours (with consultation and sample)
  Biological data obtained from lesional skin will be compared with those of healthy skin.

SECONDARY OUTCOMES:
Determination of the inflammatory profile of skin and blood during AD. Definition of the seric cytokine signature characteristic of AD. Characterization of the phenotype and function of the lymphocytic infiltrate T during AD. | 2 hours (with consultation and sample)
  Biological data obtained from lesional skin will be compared with those of healthy skin.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - CHU de Poitiers, Poitiers